CLINICAL TRIAL: NCT04191187
Title: Reduced-Intensity Fludarabine, Melphalan, and Total Body Irradiation Conditioning for Transplantation of HLA-Haploidentical Related Hematopoietic Cells (Haplo-HCT) For Patients With Hematologic Malignancies
Brief Title: Reduced Intensity Flu/Mel/TBI Conditioning for HAPLO HCT Patients With Hematologic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20131
Record Dates: First submitted 2019-12-06; First posted 2019-12-09 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Biphenotypic Acute Leukemia; Undifferentiated Leukemia; Prolymphocytic Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia; Myeloproliferative Neoplasm; Relapsed Large Cell Lymphoma; Mantle Cell Lymphoma; Hodgkin Lymphoma; Burkitt Lymphoma; Relapsed T-Cell Lymphoma; Relapsed Chronic Lymphocytic Leukemia; Relapsed Small Lymphocytic Lymphoma; Relapsed Marginal B-cell Lymphoma; Relapsed Follicular Lymphoma; Lymphoplasmacytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Biphenotypic, Acute; Leukemia, Prolymphocytic; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myeloproliferative Disorders; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Hodgkin Disease; Burkitt Lymphoma; Lymphoma, T-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone | interventions — fludarabine; fludarabine phosphate; Melphalan; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Conditioning Regimen + Transplant (Experimental): All participants will receive a conditioning regimen of Fludarabine, Melphalan and Total Body Irradiation prior to transplantation of HLA-Haploidentical Related Hematopoietic Cells (Haplo-HCT)
  Interventions: Drug: Fludarabine; Drug: Melphalan; Radiation: Total Body Irradiation

INTERVENTIONS:
Drug: Fludarabine — Fludarabine 30mg/m^2/day will be administered over 30-60 minutes intravenous infusion on Days -6 through -2 for a total dose of 150 mg/m^2
  Other Names: Fludara
Drug: Melphalan — Melphalan 70 mg/m^2 over 45 minutes will be administered Day -6. Melphalan dose will be calculated based on Actual Body Weight.
  Other Names: Alkeran
Radiation: Total Body Irradiation — Total Body Irradiation (TBI) will be delivered at a dose of 200 centigray units (cGy)

SUMMARY:
This is a single arm, phase II trial of HLA-haploidentical related hematopoietic cells transplant (Haplo-HCT) using reduced intensity conditioning (fludarabine and melphalan and total body irradiation). Peripheral blood is the donor graft source. This study is designed to estimate disease-free survival (DFS) at 18 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 55 years or HCT Co-Morbidity score (HCT-CI) >/=3
* Lack of a suitable 8/8 HLA-matched sibling donor
* Adequate performance status is defined as Karnofsky score ≥ 70%
* Patients and selected donor must be HLA typed at high resolution using DNA based typing at the following HLA-loci: HLA-A, -B, -C and DRB1. Donors must be HLA-haploidentical relatives including, but not limited to, children, siblings, or parents, defined as having a shared HLA haplotype between donor and patient at HLA-A, -B, -C, and -DRB1.
* Acute Myeloid Leukemia (AML): Must be in remission with morphology (<5% blasts)
* Acute Lymphoblastic Leukemia (ALL)/lymphoma second or greater complete remission (CR) first CR unable to tolerate consolidation chemotherapy due to chemotherapy-related toxicities, first CR high-risk ALL
* Biphenotypic/Undifferentiated/Prolymphocytic Leukemias in first or subsequent CR
* Myelodysplastic syndrome: any subtype including refractory anemia (RA) if severe pancytopenia or complex cytogenetics. Blasts must be less than 5%. If 5% of more requires chemotherapy for cytoreduction to </=5% prior to transplantation.
* Chronic Myelogenous leukemia in accelerated phase: patient must have failed at least two different Tyrosine Kinase Inhibitor (TKI)s, been intolerant to all TKIs, or have T315l mutation
* Myeloproliferative neoplasms/myelofibrosis: Blasts must be less than 5%. If 5% or more requires chemotherapy for cytoreduction to </=5% prior to transplantation
* Relapsed large-cell lymphoma, mantle-cell lymphoma or Hodgkin lymphoma that is chemotherapy sensitive and has failed or ineligible for an autologous transplant
* Burkitt's lymphoma in second CR or subsequent CR
* Relapsed T-cell lymphoma that is chemotherapy sensitive in CR/Partial Response (PR) that has failed or ineligible for an autologous transplant
* Natural killer cell malignancies
* Relapsed chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, follicular lymphoma with any of the following:
* Progressed within 12 months of achieving a partial or complete remission Patients who had remissions lasting up
* Patients who had remission lasting > 12 months are eligible after at least two prior therapies
* Patients with primary, refractory disease. Bulky disease and an estimated tumor doubling time of less than one month require debulking therapy prior to transplant.
* Lymphoplasmacytic lymphoma is eligible after initial therapy if chemotherapy sensitive
* Adequate organ function as defined per protocol
* Sexually active females of child bearing potential and males with partners of child bearing potential must agree to use adequate birth control during study treatment

Exclusion Criteria:

* Pregnant or breastfeeding
* Untreated active infection
* Active HIV infection
* Prior allogenic transplant at any time prior or less than 6 months since prior autologous transplant (if applicable)
* Active central nervous system malignancy
* Favorable risk AML defined as per protocol
* Active central nervous system malignancy
* Favorable risk AML defined as having one of the following:
* t(8,21) without cKIT mutation or evidence of immunophenotypic, cytogenetic or molecular minimal residual disease (MRD)
* inv(16) or t(16;16) without cKIT mutation or evidence of MRD
* Normal karyotype with mutated NPM1 but FLT3-ITD wild type without evidence of MRD
* Normal karyatype with double mutated CEBPA without evidence of MRD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2024-02-11 (Actual); Study Completion 2024-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelli Bejanyan, MD, Principal Investigator — Moffitt Cancer Center
Locations (1):
- H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conditioning Regimen + Transplant
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Evaluable Participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 19
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 29
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 26
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 34

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: Disease Free Survival (DFS) is defined as the time from the date of Peripheral Blood Stem Cell Transplant (PBSCT) to first documentation of relapse or death due to any cause, whichever comes first.
Time Frame: Up to 18 months post-transplant
Population: Evaluable Participants
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
percentage of participants | 70.6 [59.2 to 100]
Statistical Analysis 1: Comparison: Conditioning Regimen + Transplant; Test type: Superiority; p = 0.002, Log Rank — One sided log rank test; PFS at 18 Months = 70.8, 90% CI 1-sided [lower limit 59.2]

2. Secondary Outcome: Percentage of Participants With Graft vs Host Disease (GVHD) Free Survival
Description: GVHD-free survival is defined as the time from the date of PBSCT to date of events which include grade III-IV acute GVHD and systemic therapy-requiring chronic GVHD.
Time Frame: At 180 days post-transplant
Population: Evaluable Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
percentage of participants | 61.8 [43.4 to 75.7]

3. Secondary Outcome: Percentage of Participants Overall Survival (OS)
Description: OS is defined as the time from the date of PBSCT to the date of death due to any cause.
Time Frame: Up to 18 months
Population: Evaluable Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
percentage of participants | 73.3 [54.9 to 85.1]

4. Secondary Outcome: Percentage of Participants With Treatment Related Mortality (TRM) at 6 Months
Description: TRM is defined as death not directly due to disease
Time Frame: at 6 months post-transplant
Population: Evaluable Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
percentage of participants | 17.6 [7.0 to 32.2]

5. Secondary Outcome: Percentage of Participants With Treatment Related Mortality (TRM) at 18 Months
Description: TRM is defined as death not directly due to disease
Time Frame: at 18 months post-transplant
Population: Evaluable Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
percentage of participants | 17.6 [7.0 to 32.2]

6. Secondary Outcome: Percentage of Participants With Relapse Free Survival (RFS)
Description: RFS is defined as the time from the date of PBSCT to relapse or death.
Time Frame: Up to 18 months post-transplant
Population: Evaluable Participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Conditioning Regimen + Transplant
Number analyzed (Participants) | 34
percentage of participants | 70.6 [59.2 to 79.3]

ADVERSE EVENTS:
Time Frame: All events beginning with start of study intervention until 30 days after the last day of study intervention (up to 36 months) will be reported.
Arm/Group | Conditioning Regimen + Transplant
All-Cause Mortality (participants affected / at risk) | 9/34
Serious Adverse Events (participants affected / at risk) | 21/34
Other Adverse Events (participants affected / at risk) | 16/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conditioning Regimen + Transplant (N=34)
GVHD (Immune system disorders) | 2 (2)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 9 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
COVID-19+ (Infections and infestations) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Multi-organ failure (General disorders) | 2 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 2 (2)
Thromboembolic event (Vascular disorders) | 1 (1)
Fever (General disorders) | 5 (5)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bacteremia (Infections and infestations) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Viremia (Infections and infestations) | 2 (2)
Encephalopathy (Nervous system disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gastric hemorrhage (Gastrointestinal disorders) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 (1)
Lung Infection (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Anaphylaxis (Immune system disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 2 (3)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Encephalitis infection (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Conditioning Regimen + Transplant (N=34)
Sepsis (Infections and infestations) | 5 (6)
Cytomegalovirus infection reactivation (Infections and infestations) | 2 (2)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2)
Lung Infection (Infections and infestations) | 2 (2)
Skin Infection (Infections and infestations) | 1 (1)
Viremia (Infections and infestations) | 1 (1)
Fever (General disorders) | 4 (4)
Multi-organ failure (General disorders) | 2 (2)
Disease Progression (General disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 2 (2)
Immune system disorders - Other, specify (Immune system disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-11-22): https://cdn.clinicaltrials.gov/large-docs/87/NCT04191187/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT04191187/ICF_001.pdf